CLINICAL TRIAL: NCT02458547
Title: Effect of Anesthesia Technique on Outcome After Hip Fracture Surgery in Elderly Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4-2015-0088
Record Dates: First submitted 2015-05-26; First posted 2015-06-01 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures | interventions — Desflurane; Propofol; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group D (Experimental): General anesthesia with desflurane
  Interventions: Drug: Desflurane
- Group P (Active Comparator): General anesthesia with propofol total intravenous anesthesia
  Interventions: Drug: Propofol
- Group S (Active Comparator): Spinal anesthesia with 0.5% bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Desflurane — Inhalation anesthesia with desflurane at age-adjusted MAC of 0.8~1.0
  Arms: Group D
Drug: Propofol — Total intravenous anesthesia with propofol target controlled infusion
  Arms: Group P
Drug: Bupivacaine — Spinal anesthesia with 0.5% bupivacaine
  Arms: Group S

SUMMARY:
Despite many previous studies, whether anesthetic technique will significantly affect overall patient outcome, morbidity and mortality in elderly hip fracture patients is controversial. Due to old age, poor patient condition and emergent clinical settings, patients undergoing surgical procedures for hip fracture management are often subject to poor postoperative outcome and high mortality rates. While many studies have reported that regional anesthesia leads to improved postoperative outcome after hip fracture surgery, others have concluded otherwise. Moreover, because the majority of these previous studies are retrospective cohorts or systemic reviews, there is a need for randomized clinical trials to provide high quality evidence. This study aims to compare patient outcome between three different anesthetic techniques in elderly patients undergoing surgery for hip fracture management by evaluating proinflammatory cytokines, chemistry lab testing and clinical outcome between general anesthesia with either desflurane or propofol-based TIVA and spinal anesthesia with bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 65 years scheduled for elective or emergency hip fracture surgery.

Exclusion Criteria:

1. Patient refusal
2. Inflammation or wound at puncture site, increased intracranial pressure, bleeding diathesis
3. Allergies to propofol or its ingredients, soybeans or peanuts
4. Patients with altered mental status
5. Illiterate patients or foreigners

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 186 (Actual)
Dates: Start 2015-05; Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
HMGB1 | from preoperative baseline to 72hours
IL-6 | from preoperative baseline to 72hours
NT-proBNP | from preoperative baseline to 72hours
hemoglobin | from preoperative baseline to 72hours
total lymphocyte count | from preoperative baseline to 72hours
albumin | from preoperative baseline to 72hours
creatinine | from preoperative baseline to 72hours
potassium | from preoperative baseline to 72hours
troponin-T | from preoperative baseline to 72hours
CRP | from preoperative baseline to 72hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University Health System, Seoul, South Korea